CLINICAL TRIAL: NCT04552665
Title: Prospective Procedural Data Collection for Continuous Improvement of the KODEX - EPD™ System Performance
Acronym: KODEX
Status: Terminated | Type: Observational
Why Stopped: EPD Business was terminated
Sponsor: EPD Solutions, A Philips Company (Industry)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 20-0337
Record Dates: First submitted 2020-08-18; First posted 2020-09-17 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Cardiac Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Adults: Patients who have cardiac arrhythmia
  Interventions: Device: KODEX-EPD system

INTERVENTIONS:
Device: KODEX-EPD system — To evaluate the performance of the KODEX-EPD system and collect procedural data and medical images for Philips' internal research and development activities (R&D)

SUMMARY:
The purpose of the KODEX EPD Field study is to evaluate the performance of the KODEX-EPD system and collect procedural data and medical images for Philips' internal research and development activities (R&D) related to the KODEX-EPD system, as well as for marketing and publication purposes. The KODEX-EPD system is an imaging system that will allow for real time visualization of the catheters in your heart during your procedure, as well as display cardiac images of your heart in several different formats.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac Ablation

Exclusion Criteria:

* There is no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo a cardiac ablation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Cardiac Images | Through study completion, an average 1 year
  The KODEX-EPD system is an imaging system that will allow for real time visualization of the catheters in your heart during your procedure, as well as display cardiac images of your heart in several different formats.

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Kowalski, MD, Principal Investigator — Staten Island University Hospital North; Anneleen Viville, Study Director — EPD Solutions, A Philips Compagny
Locations (1):
- Staten Island University Hospital North Campus, Staten Island, New York, United States

IPD SHARING:
Plan to Share IPD: No